CLINICAL TRIAL: NCT02367183
Title: A Randomized, Double-blind, Multicenter Study to Explore the Effect of GED-0301 on Endoscopic and Clinical Outcomes in Subjects With Active Crohn's Disease.
Brief Title: A Randomized, Double-blind, Study to Explore the Effect of GED-0301 in Subjects With Active Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GED-0301-CD-001
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Active Crohn's Disease; GED-0301; Endoscopic; Double-Blind; IBD; Mongersen
MeSH Terms: conditions — Crohn Disease | interventions — GED0301

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GED-0301 160mg QD 12 WK (Experimental): GED-0301 160 mg once daily (QD) for 12 weeks
  Interventions: Drug: GED-0301
- GED-0301 160 mg QD 8 WK (Experimental): GED-0301 160 mg QD for 8 weeks followed by 4 weeks of placebo
  Interventions: Drug: GED-0301; Drug: Placebo
- GED-0301 160 mg QD 4 WK (Experimental): GED-0301 160 mg QD for 4 weeks followed by 8 weeks of placebo
  Interventions: Drug: GED-0301; Drug: Placebo

INTERVENTIONS:
Drug: GED-0301
Drug: Placebo
  Arms: GED-0301 160 mg QD 4 WK; GED-0301 160 mg QD 8 WK

SUMMARY:
This study is design to explore the effect of GED-0301 on clinical and endoscopic outcome and to evaluate its safety in subjects with active Crohn's disease.

DETAILED DESCRIPTION:
Approximately 51 subjects will be randomized in a 1:1:1 ratio to receive 1 of 3 treatment regimens in a 12-week Induction Phase:

GED-0301 160 mg Once Daily (QD) for 12 weeks GED-0301 160 mg Once Daily (QD) for 8 weeks followed by 4 weeks of placebo GED-0301 160 mg Once Daily (QD) for 4 weeks followed by 8 weeks of placebo Treatment assignment at baseline will be stratified via an Interactive Voice Response System (IVRS)/or an Interactive Web Response System (IWRS) based on previous exposure to TNF-α blockers (yes/no) and disease location (disease restricted to the terminal ileum and/or up to the mid transverse colon only, or disease involving at least 1 ulcerated segment distal to mid transverse colon). The number of subjects with previous exposure to TNF-α blockers is targeted to be approximately 40%. The number of subjects with disease involving distal to mid transverse colon is targeted to comprise approximately 50% of the study population.

The study will consist of 5 phases:

Screening Phase - up to 4 weeks Induction Phase - 12 weeks Eligible subjects will enter the Induction Phase at the Baseline Visit (Week 0/Induction Visit 1). Subjects will be assigned randomly to receive IP as described above.

At Induction Week 12, subjects (responders) who achieve clinical remission, defined as a CDAI score < 150, or clinical response, defined as a decrease from baseline of ≥ 100 points in Crohn's Disease Activity Index (CDAI) score, at any of the following Induction Visits (Weeks 4, 8 and/or Week 12) will enter the Observation Phase. The Observation Phase will have a duration of up to 52 weeks. Subjects who are unable to achieve clinical remission or clinical response (no responders) at the following Induction Visits (Weeks 4, 8 and Week 12), will be discontinued from the study. Subjects who enter the Observation Phase and were receiving corticosteroids at baseline will start tapering corticosteroids at the end of the Induction Phase (Induction Week 12).

Observation Phase - up to 52 weeks Subjects who enter the Observation Phase will be evaluated by CDAI score every 4 weeks. Subjects will not receive investigational product (IP) during the Observation Phase. Subjects who experience a partial loss of response or are unable to taper corticosteroids during the Observation Phase will enter the Extension Phase. Partial loss of response is defined as 2 consecutive visits with both a CDAI score ≥ 150 and an increase of CDAI score ≥ 50 points from the CDAI score at the visit when the subject was first a responder during the Induction Phase. Partial loss of response must be confirmed 2 to 4 weeks post initial identification of partial loss of response. Subjects who do not experience a partial loss of response until Observation Week 52 will have an end-of-study visit.

Extension Phase -24 weeks Subjects who enter the Extension Phase will receive GED-0301 40 mg QD on a 4-week, alternating dosing schedule (4 weeks of treatment with GED-0301, followed by 4 weeks without GED-0301 treatment) for 24 weeks.

Follow-up Phase - 4 weeks

Subjects who complete the Extension Week 24 Visit will have 2 options:

* Subjects will have the Follow-up Visit if they chose to not enter the Long-Term Extension Study or it has not been initiated
* Subjects may proceed to the Long-Term Extension Study, provided this study has been initiated by the time the subjects complete study GED-0301-CD-001 and subjects meet all inclusion/exclusion criteria of the Long-Term Extension Study.

Subjects who prematurely discontinue from the study, for any reason, will enter the Follow-up Phase, the 4-week period after the last study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female who is ≥18 years at the time of signing the Informed Consent Form (ICF).
2. Understand and voluntarily sign an Informed Consent Form (ICF) prior to conducting any study related assessments/procedures.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Diagnosis of Crohn's Disease (CD) with a duration of at least 3 months prior to screening.
5. Diagnosis of ileitis, ileocolitis or colitis , as determined by endoscopic, radiographic or any other imaging modality (eg, magnetic resonance imaging [MRI], computed tomography [CT] scan) evaluation performed within 2 years prior to screening. Subjects with colitis restricted to the left colon will not be allowed in the trial.
6. Active disease, defined as Crohn's Disease Activity Index (CDAI) score ≥ 220 and ≤ 450 (range: 0 to 600) at screening.
7. Simple Endoscopic Score for Crohn's Disease (SES-CD) score ≥ 7 at screening. Subjects with ileitis only will require Simple Endoscopic Score for Crohn's Disease (SES-CD) ≥ 4
8. Must have failed or experienced intolerance to at least one of the following:

   aminosalicylates, budesonide, systemic corticosteroids, immunosuppressants (ie, 6 mercaptopurine [6-MP], azathioprine [AZA], or methotraxate [MTX]) or tumor necrosis factor-α tumor necrosis factor-α (TNF-α) blockers (eg, infliximab, adalimumab or certolizumab) .
9. Subjects receiving oral aminosalicylates may continue their use during the study, provided that dose has been stable for at least 2 weeks prior to screening. The dose of oral aminosalicylates must remain stable through the duration of the study or early termination from the study. If oral aminosalicylates have been recently discontinued, treatment must have been stopped at least 2 weeks prior to screening.
10. Subjects receiving oral corticosteroids may continue their use during the Induction Phase, provided that the dose (prednisone ≤ 20 mg/day or equivalent, budesonide ≤ 9 mg/day) has been stable for 3 weeks prior to screening. If oral corticosteroids were recently discontinued, discontinuation must have been completed at least 4 weeks prior to screening. Corticosteroid doses should remain stable until the subject is eligible to start corticosteroids tapering.
11. Subjects receiving immunosuppressants, such as , 6 mercaptopurine (6-MP), azathioprine (AZA), or methotraxate (MTX) may continue their use during the study, provided that treatment was initiated ≥ 12 weeks prior to screening. The dose of immunosuppressants must be at a stable dose for ≥ 8 weeks prior to the Baseline Visit and must remain stable through the duration of the study or early termination from the study. Subjects who discontinued immunosuppressants should have stopped them at least 8 weeks prior to screening.
12. Must meet the following laboratory criteria:

    1. White blood cell count ≥ 3000/mm3 (≥ 3.0 X 10^9//L) and < 14,000/mm3 (< 14.0 X 10^9/L)
    2. Platelet count ≥ 100,000/mm3 (≥ 100 X 10^9/L)
    3. Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
    4. Aspartate aminotransferase (AST) / serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) / serum glutamic-pyruvic transaminase (SGPT) ≤ 2 X upper limit of normal (ULN)
    5. Total bilirubin ≤ 2 mg/dL (≤ 34 μmol/L) unless there is a confirmed diagnosis of Gilbert's disease
    6. Hemoglobin ≥ 9 g/dL (≥ 5.6 mmol/L)
    7. Activated partial thromboplastin time (APTT) ≤ 1.5 X ULN
13. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and the Baseline Visit. While on IP and for at least 28 days after the Early Termination Visit or the end-of-study visit (Observation Week 52 or Extension Week 24), FCBP who engage in activity in which conception is possible must use 1 of the approved contraceptive options2 described below: Option 1: Any one of the following highly effective methods: hormonal contraception (for example, birth control pills, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation (tying your tubes); or a partner with a vasectomy OR

    Option 2: Any two of the following effective methods: male or female condom PLUS one of the following additional barrier methods:
    1. diaphragm with spermicide;
    2. cervical cap with spermicide; or
    3. contraceptive sponge with spermicide
14. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on Investigational Product (IP) and for at least 28 days after the Early Termination Visit or the end-of-study visit (Observation Week 52 or Extension Week 24).

Exclusion Criteria:

1. Diagnosis of Crohn's colitis restricted to the left colon , ulcerative colitis (UC), indeterminate colitis, ischemic colitis, microscopic colitis, radiation colitis or diverticular disease-associated colitis.
2. Local manifestations of Crohn's Disease (CD) such as strictures, abscesses, fistula, short bowel syndrome or other disease complications for which surgery might be indicated or could confound the evaluation of efficacy.
3. Intestinal resection within 6 months or any intra-abdominal surgery within 3 months prior to screening.
4. Subjects with an ileostomy or a colostomy.
5. Stool positive for any enteric pathogen or C. difficile toxin at screening.
6. History of colorectal cancer or colorectal dysplasia.
7. Prior use of mycophenolic acid, tacrolimus, sirolimus, cyclosporine, thalidomide or apheresis (eg, Adacolumn) for the treatment of CD. In addition, prior use of any of these treatment modalities for an indication other than CD within 8 weeks of screening is also excluded.
8. Use of intravenous (IV) corticosteroids within 2 weeks of screening.
9. Use of topical treatment with 5 aminosalicylic acid (5-ASA) or corticosteroid enemas or suppositories within 2 weeks of screening
10. Use of antibiotic therapy for the treatment of Crohn's Disease (CD) within 3 weeks of screening.
11. Use of cholestyramine within 3 weeks of screening.
12. Prior treatment with more than 2 tumor necrosis factor-α (TNF-α) blockers.
13. Prior treatment with any integrin antagonists (eg, natalizumab or vedolizumab).
14. Use of tumor necrosis factor-α (TNF-α) blockers within 12 weeks of the screening
15. Administration of total parenteral nutrition (TPN) within 4 weeks of screening.
16. History of any clinically significant neurological, renal, hepatic, gastrointestinal, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, or any other medical condition that, in the Investigator's opinion, would prevent the subject from participation in the study.
17. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she was to participate in the study or confounds the ability to interpret data from the study.
18. Pregnant or breastfeeding.
19. History of any of the following cardiac conditions within 6 months of screening: myocardial infarction, acute coronary syndrome, unstable angina, new onset atrial fibrillation, new onset atrial flutter, second- or third-degree atrioventricular block, ventricular fibrillation, ventricular tachycardia, heart failure, cardiac surgery, interventional cardiac catheterization (with or without a stent placement), interventional electrophysiology procedure, or presence of implanted defibrillator.
20. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease and Herpes zoster), human immunodeficiency virus (HIV), or any major episode of infection requiring hospitalization or treatment with intravenous (IV) or oral antibiotics within 4 weeks of screening.
21. History of congenital or acquired immunodeficiency (eg, common variable immunodeficiency disease).
22. History of malignancy, except for:

    1. Treated (ie, cured) basal cell or squamous cell in situ skin carcinomas
    2. Treated (ie, cured) cervical intraepithelial neoplasia or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years
23. Subjects who have received any investigational drug or device within 1 months of screening.
24. Prior treatment with GED-0301, or participation in a clinical study involving GED-0301.
25. History of alcohol, drug, or chemical abuse within the 6 months prior to screening.
26. Known hypersensitivity to oligonucleotides or any ingredient in the IP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Change in SES-CD Score | Week 12
  The change from baseline in the Simplified Endoscopic Activity Score for Crohn's disease (SES-CD) score at Induction Week 12.

SECONDARY OUTCOMES:
Proportion of subjects achieving a clinical remission, defined as a CDAI score < 150 at Induction Week 4 | Week 4
  Clinical remission is defined as a Crohn's Disease Activity Index (CDAI) score < 150
Adverse Event (AE) | Up to 97 weeks
  Assessed by the type, frequency and severity of adverse events, and its relationship to investigational product (IP), discontinuation due to adverse events, and clinically significant changes in vital signs, Electrocardiograms (ECGs), and/or laboratory findings.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Rossiter, MD, Study Director — Celgene
Locations (50):
- United States (34):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Macks Research Group, Newport Beach, California
  - Medical Associates Research Group, San Diego, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Florida Research Network, LLC, Gainesville, Florida
  - University of Florida Shands Endoscopy Center University of Florida at Gainesville, Gainesville, Florida
  - Borland - Groover Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Gastroenterology Specialists, Suwanee, Georgia
  - University of Louisville, Louisville, Kentucky
  - Metropolitan Gastroenterology, Chevy Chase, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Concorde Medical Group, New York, New York
  - Cornell University, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cumberland Research Associates, Fayetteville, North Carolina
  - The Management Associates, Wilmington, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Nashville Gastrointestinal Specialists, Nashville, Tennessee
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - Digestive Disease Consultants, Grapevine, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Digestive Disease Consultants - Southlake, Irving, Texas
  - University of Utah Division of Gastroenterology, Salt Lake City, Utah
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Australia (5):
  - Centre For Digestive Diseases, Five Dock, New South Wales
  - Mater Adult Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Concord Repatriation General Hospital, Concord
- Canada (4):
  - GI Research Institute, Vancouver, British Columbia
  - PerCuro Clinical Research, Victoria, British Columbia
  - London Health Science Center U. Hospital, London, Ontario
  - McMaster University Medical Centre, West Hamilton, Ontario
- Hungary (2):
  - Szent Imre Korhaz, Budapest
  - Szegedi Tudomanyegyetem, Szeged
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Bratislava
  - IBD Centrum s.r.o., Bratislava
  - KM Management, spol. s r.o., Nitra
  - GASTRO I., s.r.o., Prešov

REFERENCES:
- [Derived] Feagan BG, Sands BE, Rossiter G, Li X, Usiskin K, Zhan X, Colombel JF. Effects of Mongersen (GED-0301) on Endoscopic and Clinical Outcomes in Patients With Active Crohn's Disease. Gastroenterology. 2018 Jan;154(1):61-64.e6. doi: 10.1053/j.gastro.2017.08.035. Epub 2017 Aug 25. PMID 28847751